CLINICAL TRIAL: NCT04461145
Title: Effect of Dual Tasks on Gait Symmetry After Anterior Cruciate Ligament Reconstruction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: OR002
Record Dates: First submitted 2020-06-29; First posted 2020-07-08 (Actual); Last update posted 2020-07-08 (Actual); Status verified 2020-06

CONDITIONS: Anterior Cruciate Ligament Injury
Keywords: anterior cruciate ligament; knee; biomechanics; walking; cognition
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ACL group (Other)
  Interventions: Behavioral: command

INTERVENTIONS:
Behavioral: command — The participant was asked to walk along the walkway while backward counting numbers with increment of seven starting from a randomly given number.

SUMMARY:
Individuals who received anterior cruciate ligament (ACL) reconstruction demonstrated lower extremity movement asymmetries. The purpose of this study was to determine if psychological impairment was a contributor to lower extremity movement asymmetries in walking for individuals who received ACL reconstruction.

DETAILED DESCRIPTION:
Background: Anterior cruciate ligament (ACL) reconstruction is a commonly surgical procedure to restore knee functions after an ACL injury. Lower extremity movement asymmetries were found to be predictive of ACL re-injury and knee OA after ACL reconstruction. Although these studies indicated that psychological impairments may contribute to patients' movement asymmetries after ACL reconstruction surgery, the effect of psychological impairment on lower extremity movement asymmetries has not been confirmed yet.

Methods: Each participant was asked to wear a pair of black spandex shorts. Passive reflective markers were placed bilaterally at the anterior superior iliac spine, posterior superior iliac spine, lateral thigh, lateral femoral condyle, medial femoral condyle, anterior superior shank, anterior inferior shank, lateral malleoli, medial malleoli, heel, and first and fifth metatarsophalangeal. The participant was instructed to walk with barefoot in two conditions: (1) without cognitive task (single-task condition), and (2) with concurrent cognitive task (dual-task condition). In single-task condition, the participant walked along a 10-m walkway at self-selected walking speed. In dual-task condition, the participant walked along the walkway while backward counting numbers with an increment of seven starting from a randomly given number between 125 and 250. In dual-task condition, participants immediately initiated the walking task at their preferred speed once they heard the number read by the investigator and kept counting out loudly as required without repeating the given number. Participants were asked to count as fast as possible while walking task. A 5 min rest was requested between single-task and dual-task test. The order of conditions was randomized for the participant. Quadriceps strength was evaluated for the participant after walking test.

Three-dimensional (3-D) trajectories of the reflective markers were collected using an 8-camera motion capture system (VICON, Oxford, UK) at a sample rate of 100 Hz. Ground-reaction force signals were collected using two embedded force plates (AMTI, Watertown, Massachusetts) at a sample rate of 1000 Hz. Each participant was asked to have three successful trials for each condition. A successful trial was defined as a trial in which the participant performed the task as required, and all kinematic and kinetic data were collected.

Quadriceps isometric strength was quantified with an isokinetic dynamometer (CON-TREX MJ; Germany) during a maximum voluntary isometric contraction (MVIC). The participant was seated with a hip flexed at 90° and knee flexed at 60°. The lateral femoral condyle was aligned with the dynamometer axis, and the dynamometer resistance pad was secured to the anterior aspect of the distal shank. After correcting for leg weight, the participant was asked to perform submaximal practice to familiarize themselves with the testing apparatus. After familiarization of testing apparatus, the participant was asked to have three recorded maximum-effort trials (5 seconds in duration, 60 seconds' rest between trials) for each leg with uninjured leg tested first.

ELIGIBILITY:
Inclusion Criteria:

* 18-40 years old
* received unilateral ACL reconstruction

Exclusion Criteria:

* combined with other ligament injuries
* moderate or severe articular cartilage damage to the patellofemoral and tibiofemoral joint
* combined with meniscus injuries that needed to be repaired with a resection or suture
* other current orthopaedic injuries or disorders that were still affecting lower extremity movements

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2016-11-08 (Actual); Primary Completion 2017-10-20 (Actual); Study Completion 2017-10-31 (Actual)

PRIMARY OUTCOMES:
knee joint angles | at 6 months after the surgery.
  Three-dimensional gait analysis system were used during walking.
the moment of knee flexion in the gait cycle | at 6 months after the surgery.
  Three-dimensional gait analysis system were used during walking.
the moment of knee extension in the gait cycle | at 6 months after the surgery.
  Three-dimensional gait analysis system were used during walking.

SECONDARY OUTCOMES:
quadriceps strength | at 6 months after the surgery.
  Isokinetic muscle strength testing instrument were used to evaluate musle strength.
walking speed | at 6 months after the surgery.
  Three-dimensional gait analysis system were used during walking.
The International Knee Documentation Committee (IKDC) score | at 6 months after the surgery.
  The International Knee Documentation Committee (IKDC) score was used to evaluate the knee health.The patients completed score by themselves. The lowest score is 0 and the highest score is 100.

CONTACTS AND LOCATIONS:
Overall Officials: Hongshi Huang, Doctor, Study Chair — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No